CLINICAL TRIAL: NCT03391700
Title: Effect of Intraoperative Muscle Relaxation Depth on Postoperative Sore Throat and Hoarseness After General Anesthesia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: SMG-SNU Boramae Medical Center (Other)
Responsible Party: Principal Investigator, Jin-Young Hwang, associate professor, SMG-SNU Boramae Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 20170601/10-2017-4/071
Record Dates: First submitted 2017-11-09; First posted 2018-01-05 (Actual); Last update posted 2018-06-26 (Actual); Status verified 2018-06

CONDITIONS: Sore Throat
Keywords: muscle relaxant
MeSH Terms: conditions — Pharyngitis; Muscle Hypotonia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Moderate muscle relaxation (Active Comparator): Rocuronium is administered to maintain moderate relaxation during operation. This is conventional muscle relaxation level of this institute.
  Interventions: Drug: Rocuronium(moderate)
- Deep muscle relaxation (Experimental): Rocuronium is administered to maintain deep relaxation during operation.
  Interventions: Drug: Rocuronium(deep)

INTERVENTIONS:
Drug: Rocuronium(deep) — In the group with deep relaxation during surgery, rocuronium is given by continuous infusion (0.6 mg/kg/h).
  Arms: Deep muscle relaxation
Drug: Rocuronium(moderate) — In the group with deep relaxation during surgery, rocuronium is given by bolus dose(0.15mg/kg) induced a train of four count of 1-2.
  Arms: Moderate muscle relaxation

SUMMARY:
Investigators assess and compare postoperative sore throat and hoarseness in the group maintaining moderate relaxation and deep relaxation during operation.

DETAILED DESCRIPTION:
In this sturdy, the deep block is applied when the surgeon requests for deep muscle relaxation to improve surgical field condition in the surgery such as laparotomy known that the deep block is helpful and in the other surgeries, the moderate block is maintained. The investigators assess the postoperative sore throat and hoarseness and compare the effect of muscle relaxation depth in the deep block group and moderate block group in terms of the incidence and severity of postoperative sore throat and hoarseness.

ELIGIBILITY:
Inclusion Criteria:

* Requirement for mechanical ventilation under general anesthesia

Exclusion Criteria:

* Hoarseness and sore throat existed before surgery
* Upper respiratory infection
* Known or predicted difficult airway
* Liver, renal disease
* Requirement of postoperative ventilator care
* the operation within 2hrs
* Laparoscopic surgery
* Other positions except supine during surgery

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 206 (Estimated)
Dates: Start 2017-08-01 (Actual); Primary Completion 2018-07-14 (Estimated); Study Completion 2019-08-14 (Estimated)

PRIMARY OUTCOMES:
Overall incidence of postoperative sore throat | Within 24 hrs after operation
  The overall cumulative incidence of postoperative sore throat is assessed in the 24-hr evaluation period

SECONDARY OUTCOMES:
The incidence of postoperative sore throat | At 1,6, and 24 hrs after operation
  The presence of sore throat is assessed.
The severity of postoperative sore throat | At 1,6, and 24 hrs after operation
  The severity of sore throat is assessed by using a 100-point numerical ratig scale (NRS, 0 [no pain], 100 [worst pain imaginable]).
Incidence and severity of postoperative hoarseness | At 1,6, and 24 hrs after operation
  Hoarseness is defined as a voice quality different from the preoperative voice and graded as follows: none (no hoarseness), mild (recognized by the patient), moderate (obvious to the investigator), and severe (aphonia).
Postoperative analgesic consumption | Within 24 hrs after operation
  The amount of patient-controlled analgesia and other analgesic medication used

CONTACTS AND LOCATIONS:
Overall Officials: Jee-eun Chang, M.D, Principal Investigator — SMG-SNU Boramae Medical Center
Locations (1):
- Jee-Eun Chang, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No